CLINICAL TRIAL: NCT00678912
Title: Single Center Randomized Clinical Trial Comparing Weaning From Mechanical Ventilation With Computer-driven System vs Usual Care in Children
Brief Title: Weaning Children From Mechanical Ventilation:Computer-driven System Versus Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Philippe Jouvet, Associate Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUSJ-2239
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; automated weaning; children
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Children are mechanically ventilated with Smartcare/PS
  Interventions: Device: Smartcare/PS
- 2 (No Intervention): Children are mechanically ventilated with usual care

INTERVENTIONS:
Device: Smartcare/PS — computer-driven protocol that adjusts pressure support level in pressure support mode to patient respiratory status
  Other Names: Weaning from mechanical ventilation with Smartcare/PS
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether a computer-driven system (Smartcare/PS) decreases weaning duration from mechanical ventilation when compared to usual care in children.

DETAILED DESCRIPTION:
Baseline data: All subjects included into this RCT will undergo routine examination upon admission to the hospital. These examinations include physical, medical/medication history (on the last year for medical history and the last 3 months for medication history (if available), vital signs, radiologic data and laboratory tests.

Intervention: A pre-inclusion test (pressure support test) with a level of pressure support of ± 5 cmH2O of the P plateau, but no greater than 30 cmH2O (pressure-support level plus positive end-expiratory pressure), is performed to evaluate the patient's tolerance of this ventilation mode; the test is repeated daily until positive. The test could be stopped before 30 minutes if the patient showed evidence of respiratory distress (respiratory rate > 40 breaths per minute and FiO2 > 60% in order to obtain pulse oxymetry ≥ 95%). The test is considered positive when, after 30 minutes, the patient remained clinically stable with a respiratory rate lower than 40 breaths per minute and an expiratory tidal volume higher than 6 ml per kilogram of body weight within the authorized pressure-support range, with pulse oxymetry no lower than 95 percent when the fraction of inspired oxygen was no greater than 60 percent. When the pressure-support test is positive, the patient is randomized either to Arm 1 where the intervention is weaning with the support of Smartcare/PS or to Arm 2 where the intervention is weaning based on usual care. Both group are ventilated with the same ventilator: Evita XL.

ELIGIBILITY:
Inclusion Criteria:

* The attending physician thinks that the patient will be able to breathe spontaneously or the patients is already breathing spontaneously.
* No vasopressor or inotropic medication, unless the patient is receiving some digitalin or small doses of dopamine (< 5 µg/kg/min)
* Slight or no endotracheal tube gas-leakage ([Vti - Vte]/Vti ≤ 20%)
* Mechanical ventilation with a plateau pressure ≤ 25 cmH2O over PEEP
* PEEP ≤ 8 cmH2O
* FiO2 ≤ 60% in order to obtain pulse oxymetry ≥ 95%
* PaCO2 < 70 mmHg on the last blood gases
* Extubation not expected the day of inclusion

Exclusion Criteria:

* N/A

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Length of weaning from mechanical ventilation that corresponds to the time from Time 0 to the first extubation. | first extubation or 28 days

SECONDARY OUTCOMES:
Total mechanical ventilation duration | first extubation or 28 days
Proportion of time in the acceptable breathing zone | first extubation or 28 days
Weaning failure | 48 hours after first extubation
Number of interventions on the ventilator by a physician or physiotherapist | First extubation or 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Jouvet, MD PhD, Principal Investigator — Université de Montreal
Locations (1):
- CHU Sainte Justine, Montreal, Quebec, Canada

REFERENCES:
- [Background] Jouvet P, Farges C, Hatzakis G, Monir A, Lesage F, Dupic L, Brochard L, Hubert P. Weaning children from mechanical ventilation with a computer-driven system (closed-loop protocol): a pilot study. Pediatr Crit Care Med. 2007 Sep;8(5):425-32. doi: 10.1097/01.PCC.0000282157.77811.F9. PMID 17693913
- [Derived] Jouvet PA, Payen V, Gauvin F, Emeriaud G, Lacroix J. Weaning children from mechanical ventilation with a computer-driven protocol: a pilot trial. Intensive Care Med. 2013 May;39(5):919-25. doi: 10.1007/s00134-013-2837-8. Epub 2013 Jan 30. PMID 23361631